CLINICAL TRIAL: NCT02299479
Title: Adjusting Insulin Delivery to Activity (AIDA)
Brief Title: Adjusting Insulin Delivery to Activity
Acronym: AIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael Agus, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-P00014511
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Diabetes; Nocturnal Hypoglycemia
Keywords: insulin pump; continuous glucose monitor; activity monitor
MeSH Terms: conditions — Diabetes Mellitus | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Volunteers will wear a Dexcom G4 Platinum CGM device as well as an activity monitor. Data will be uploaded to study investigators on a regular basis, and recommendations will be made to adjust insulin dosing based upon analysis of these data.
  Interventions: Device: Dexcom G4 Platinum CGM; Device: Activity monitor

INTERVENTIONS:
Device: Dexcom G4 Platinum CGM — Blood glucose levels will be monitored using continuous glucose monitors (CGMs). Participants will be asked to verify CGM low blood sugars using their home glucometer. Insulin dose adjustments will be made if there is concern that nocturnal hypoglycemia is occurring in relation to high daytime activity.
  Other Names: Continuous glucose monitor and activity monitor
Device: Activity monitor — Participants will be asked to wear an activity monitor so that we may assess their daily activity level. Insulin dose adjustments will be made if there is concern that nocturnal hypoglycemia is occurring in relation to high daytime activity.

SUMMARY:
Increased daytime activity in children and adolescents with type I diabetes is known to be associated with overnight hypoglycemia. We therefore wish to perform a prospective clinical study to assess the feasibility of using activity monitor data to adjust insulin pump basal rates and see whether we can help prevent overnight hypoglycemia or decrease related interventions following high activity days. We plan to carry this out by enrolling 20 subjects (10 subjects 1 to <7 years old and 10 subjects 7 to 17 years old) with type 1 diabetes managed on insulin pump therapy and having them wear activity monitors and CGMs for up to 3 months. After an initial two-week period to establish activity baselines, we will recommend nighttime basal insulin rate adjustments based on activity monitor, CGM and insulin pump data.

DETAILED DESCRIPTION:
This study is a pilot trial investigating the feasibility of using activity monitoring data to adjust insulin pump therapy and prevent hypoglycemia. The study will enroll 20 patients with type 1 diabetes mellitus on insulin pump therapy, 10 from each of two age groups: younger children aged 1 year to <7 years of age, and older children aged 7-17 years of age. Subjects will be provided with continuous glucose monitors (DexCom G4) and activity monitors. Study duration will be up to 3 months. During the course of the study patients will continue to receive routine care by their primary endocrinologist and diabetes nurse educator (DNE). Insulin dose adjustments unrelated to activity monitor data will continue to be at the discretion of the patient's primary diabetes team.

Activity level (steps and calories burned) will be uploaded over the web in a secure fashion to our central firewall-protected database on a daily basis while CGM glucose values and insulin pump data will be collected once a week. The initial 2 weeks of a subject's enrollment in the study will be used to establish his or her baseline activity level and no changes to the insulin regimen will be made based on the activity monitor data. During weeks 3 to 12, activity data will be reviewed daily and an alternate basal insulin rate will be recommended on days considered to be increased activity days. We will use an adaptive algorithm to help guide suggested insulin basal rate changes. All recommendations will be reviewed and approved by a physician prior to implementation. The alternate rate will be derived using the subject's usual care pump settings as an initial starting point from which to make incremental changes in the 3 hour interval leading up to the hypoglycemic event. Target will be the overnight nadir obtained with usual care settings. Residual error (CGM-target) will be used to assess the validity of using the 3 hour window prior to the event to effect lower basal.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes (as clinically diagnosed by outpatient endocrinologist).
* Treated with insulin pump therapy for greater than or equal 6 months
* HbA1C of <8.5% in the previous 3 months
* Families will need to have access to Wi-Fi and a compatible smartphone in order for the data from the activity monitor and other devices to be transmitted to the research team

Exclusion Criteria:

• Current oral steroid use or other medication known to affect insulin action at investigator's discretion.

***Note: currently only enrolling patients followed at Boston Children's Hospital

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Agus, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Agus MS, Asaro LA, Steil GM, Alexander JL, Silverman M, Wypij D, Gaies MG; SPECS Investigators. Tight glycemic control after pediatric cardiac surgery in high-risk patient populations: a secondary analysis of the safe pediatric euglycemia after cardiac surgery trial. Circulation. 2014 Jun 3;129(22):2297-304. doi: 10.1161/CIRCULATIONAHA.113.008124. Epub 2014 Mar 26. PMID 24671945
- [Background] Steil GM. Algorithms for a closed-loop artificial pancreas: the case for proportional-integral-derivative control. J Diabetes Sci Technol. 2013 Nov 1;7(6):1621-31. doi: 10.1177/193229681300700623. PMID 24351189
- [Background] Agus MS, Steil GM, Wypij D, Costello JM, Laussen PC, Langer M, Alexander JL, Scoppettuolo LA, Pigula FA, Charpie JR, Ohye RG, Gaies MG; SPECS Study Investigators. Tight glycemic control versus standard care after pediatric cardiac surgery. N Engl J Med. 2012 Sep 27;367(13):1208-19. doi: 10.1056/NEJMoa1206044. Epub 2012 Sep 7. PMID 22957521
- [Background] Dauber A, Corcia L, Safer J, Agus MS, Einis S, Steil GM. Closed-loop insulin therapy improves glycemic control in children aged <7 years: a randomized controlled trial. Diabetes Care. 2013 Feb;36(2):222-7. doi: 10.2337/dc12-1079. Epub 2012 Oct 1. PMID 23033237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty participants aged 1 to 17 years were recruited at Boston Children's Hospital beginning in July of 2015.
Groups:
- Dexcom G4 Platinum CGM & Activity Monitor: Volunteers will wear a Dexcom G4 Platinum CGM device as well as an activity monitor. Data will be uploaded to study investigators on a regular basis, and recommendations will be made to adjust insulin dosing based upon analysis of these data.
  Dexcom G4 Platinum CGM: Blood glucose levels will be monitored using continuous glucose monitors (CGMs). Participants will be asked to verify CGM low blood sugars using their home glucometer. Insulin dose adjustments will be made if there is concern that nocturnal hypoglycemia is occurring in relation to high daytime activity.
  Activity monitor: Participants will be asked to wear an activity monitor so that we may assess their daily activity level. Insulin dose adjustments will be made if there is concern that nocturnal hypoglycemia is occurring in relation to high daytime activity.
Period: Overall Study
Arm/Group | Dexcom G4 Platinum CGM & Activity Monitor
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Dexcom G4 Platinum CGM and Activity Monitor: Volunteers will wear a Dexcom G4 Platinum CGM device as well as an activity monitor. Data will be uploaded to study investigators on a regular basis, and recommendations will be made to adjust insulin dosing based upon analysis of these data.
  Dexcom G4 Platinum CGM: Blood glucose levels will be monitored using continuous glucose monitors (CGMs). Participants will be asked to verify CGM low blood sugars using their home glucometer. Insulin dose adjustments will be made if there is concern that nocturnal hypoglycemia is occurring in relation to high daytime activity.
  Activity monitor: Participants will be asked to wear an activity monitor so that we may assess their daily activity level. Insulin dose adjustments will be made if there is concern that nocturnal hypoglycemia is occurring in relation to high daytime activity.
Arm/Group | Dexcom G4 Platinum CGM and Activity Monitor
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: Years] | 12 [7 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 18.7 (0.6)
Total Daily Insulin Use [Median (Full Range); unit: units of insulin/kg/day] | 0.8 [0.55 to 1.12]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Supplemental Carbohydrate Interventions up to 3 Months From Baseline.
Description: Median and inter-quartile range (IQR) of supplemental carbohydrate (SC) interventions (number of SC given by parent divided by the number of days the SC were given) to prevent hypoglycemia during the study period will be compared to those given during the baseline period for each subject. The median and IQR of all subjects will then be calculated.
Time Frame: Up to 3 months
Measure: Median (Inter-Quartile Range); unit: Supplemental Carb (SC) admin. per night
Arm/Group | Dexcom G4 Platinum CGM & Activity Monitor
Number analyzed (Participants) | 18
Supplemental Carb (SC) admin. per night | 0.11 [0.00 to 0.16]

2. Secondary Outcome: Correlation of Daytime Activity With Nighttime Nadir Glucose.
Description: Daytime activity will be determined based on steps and calories burned measured by activity monitor. High activity is defined as activity level more than 2 standard deviations above the subject's baseline. Correlations will be performed to assess if there is relationship between daytime activity (8 am to 9 pm) and nighttime nadir blood glucose level (mg/dL).
Time Frame: Up to 3 months
Measure: Median (Inter-Quartile Range); unit: Correlation coefficient
Arm/Group | Dexcom G4 Platinum CGM & Activity Monitor
Number analyzed (Participants) | 18
Correlation coefficient | 0.10 [0.01 to 0.27]

3. Secondary Outcome: Change From Baseline in Supplemental Carbohydrate Interventions up to 3 Months From Baseline in Subjects With Activity Effect.
Description: For subjects with an activity effect (subjects with a correlation between daytime activity and nighttime nadir glucose), median and inter-quartile range (IQR) of supplemental carbohydrate (SC) interventions (number of SC given by parent divided by the number of nights the SC were given) to prevent hypoglycemia during the study period will be compared to those given during the baseline period for each subject. The median and IQR of this subset of subjects will then be calculated.
Time Frame: Up to 3 months
Measure: Median (Inter-Quartile Range); unit: Carbohydrate interventions per night
Arm/Group | Dexcom G4 Platinum CGM & Activity Monitor
Number analyzed (Participants) | 10
Carbohydrate interventions per night | 0 [0 to 0.16]

ADVERSE EVENTS:
Time Frame: Entire course of the protocol, up to 3 months
Arm/Group | Dexcom G4 Platinum CGM & Activity Monitor
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexcom G4 Platinum CGM & Activity Monitor (N=20)
Medication Error (mother incorrectly programmed insulin pump) (Endocrine disorders) | 1 (1) — Mother found patient to be hyperglycemic, called clinician. Determined she had incorrectly programmed the insulin pump, patient was treated. Hyperglycemia and ketosis resolved within three hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT02299479/Prot_SAP_000.pdf